CLINICAL TRIAL: NCT04467164
Title: Vagus Nerve Stimulation: Integration of Behavior and Cardiac Modulation
Acronym: tVNS-MDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jill M. Goldstein, Ph.D., Professor & Exec. Dir. Innovation Center on Sex Differences in Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2013P001259; R21MH103468 (NIH)
Record Dates: First submitted 2020-07-01; First posted 2020-07-10 (Actual); Results first posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Major Depressive Disorder
Keywords: Transcutaneous vagus nerve stimulation; Stress response circuitry; functional magnetic resonance imaging; respiration; depression
MeSH Terms: conditions — Depressive Disorder, Major; Respiratory Aspiration; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exhalatory-gated tVNS (Experimental): exhalatory-gated tVNS on the left auricle
  Interventions: Other: exhalatory-gated transcutaneous vagus nerve stimulation (e-RAVANS)
- Inhalatory-gated tVNS (Active Comparator): inhalatory-gated tVNS on the left auricle
  Interventions: Other: Inhalatory-gated transcutaneous vagus nerve stimulation (i-RAVANS)

INTERVENTIONS:
Other: exhalatory-gated transcutaneous vagus nerve stimulation (e-RAVANS) — Non-painful exhalatory-gated electrical stimulation of the auricle for 30 minutes during a functional magnetic resonance imaging session.
  Other Names: e-RAVANS
  Arms: Exhalatory-gated tVNS
Other: Inhalatory-gated transcutaneous vagus nerve stimulation (i-RAVANS) — Non-painful inhalatory-gated electrical stimulation of the auricle for 30 minutes during a functional magnetic resonance imaging session.
  Other Names: i-RAVANS
  Arms: Inhalatory-gated tVNS

SUMMARY:
This study characterized the impact of respiratory-gated transcutaneous vagus nerve stimulation (tVNS) on the modulation of the stress response circuitry, vagal tone and depressed mood in patients with major depressive disorder (MDD). Twenty premenopausal women with recurrent MDD in an active episode were recruited into a single-blind cross-over study that included two functional MRI visits within a one week period with simultaneous mood and physiological assessments. Randomization to exhalatory- or inhalatory-gated tVNS was performed to control for order effects. The study hypothesis was that exhalatory-gated tVNS would have a significantly greater impact on the regulation of brain activity in stress response circuitry, vagal tone and depressed mood in MDD patients compared to inhalation-gated tVNS. This is not a clinical trial aimed to test a medical device, but a basic experimental study oriented to understand the effects of vagal afference modulation on brain and cardiovagal physiological response to stress in major depression.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) has been associated with alterations of the stress response circuitry, including the hypothalamus, amygdala, hippocampus, anterior cingulate cortex, ventromedial, dorsolateral and orbital prefrontal cortices. Many of these regions are morphologically and functionally sexually dimorphic and associated with vulnerability for sex differences in MDD. A major role for the stress response circuitry is to assess potentially stressful stimuli and respond with a neuroendocrine signal that coordinates homeostatic responses throughout the body. Neuroimaging studies have suggested that alterations in this circuitry are implicated in mood dysregulation, increased activation of the hypothalamic-pituitary-adrenal (HPA) axis, and imbalance between the sympathetic and parasympathetic nervous system in depressed persons. A better understanding of the mechanisms underlying alterations in physiological response to stress in major depression may contribute to the development of novel interventions that regulate this system with a significant impact on the improvement of clinical and physiological alterations of MDD.

It has been previously suggested that modulation of vagus nerve activity may have a significant effect on the modulation of the brain circuitry involved in the regulation of mood and stress response. Recently, a non-invasive approach for modulation of vagus nerve activity, transcutaneous auricular vagus nerve stimulation (tVNS), which targets the auricular branch of the vagus nerve (ABVN) has been proposed. Moreover, previous studies have shown that vagal afference is highly regulated by respiration and that modulation of vagus nerve activity may be optimized by gating ABVN stimulation to the exhalatory phase of the respiratory cycle. Thus, this study proposed to characterize the impact of respiratory-gated tVNS on the modulation of the stress response circuitry, vagal tone and depressed mood in patients with recurrent major depression (MDD). This is not a clinical trial aimed to test a medical device, but a basic experimental study oriented to understand the effects of vagal afference modulation on brain and cardiovagal physiological response to stress in major depression.

Twenty premenopausal women with recurrent MDD in an active episode were recruited into a single-blind cross-over study that included two functional MRI visits, within a one week period, with simultaneous mood and physiological assessments. Randomization to exhalatory- or inhalatory-gated tVNS was performed to control for order effects. Subjects were exposed to a mild visual stress challenge that preceded and followed 30 minutes of exhalatory- or inhalatory-gated tVNS. The study hypothesis was that exhalatory-gated tVNS would have a significantly greater impact on the regulation of brain activity in stress response circuitry, vagal tone and depressed mood in MDD patients compared to inhalation-gated tVNS

ELIGIBILITY:
Inclusion Criteria: Recurrent MDD diagnosis (≥ 2 episodes) with a current active depressive episode.

Exclusion Criteria:

* History of Axis I psychiatric diagnosis other than MDD or anxiety disorder - e.g., substance use disorder, psychotic disorder, or bipolar disorder.
* Current Suicidal Ideation with intent and/or plan or history of suicide attempt within the last year
* Use of psychotropic medications within four weeks prior to study with the exception of Selective Serotonin Reuptake Inhibitors (SSRIs) and Selective Norepinephrine Reuptake Inhibitors (SNRIs) class of antidepressant medication only
* Use of Tricyclic antidepressants (TCAs), Monoamine oxidase inhibitors (MAOIs), and Atypical agents
* History of cardiovascular disease
* History of neuroleptic use
* Past history of substance abuse or dependence within the past 12 months (excludes nicotine)
* Bleeding disorder or use of anticoagulants.
* Pregnancy
* Metallic implants or devices contraindicating magnetic resonance imaging.
* Use of beta blockers

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — premenopausal women only
Enrollment: 20 (Actual)
Dates: Start 2015-04-15 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill M Goldstein, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Exhalatory-gated tVNS Then Inhalatory-gated tVNS: Participants first received exhalatory-gated tVNS for 30 minutes during a first functional MRI session. After a washout period of 1 week, they then received inhalatory-gated tVNS for 30 minutes during a second fMRI session.
- Inhalatory-gated tVNS Then Exhalatory-gated tVNS: Participants first received inhalatory-gated tVNS for 30 minutes during a first functional MRI session. After a washout period of 1 week, they then received exhalatory-gated tVNS for 30 minutes during a second fMRI session.
Period: First Intervention (30 Minutes)
Arm/Group | Exhalatory-gated tVNS Then Inhalatory-gated tVNS | Inhalatory-gated tVNS Then Exhalatory-gated tVNS
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Washout (1 Week)
Arm/Group | Exhalatory-gated tVNS Then Inhalatory-gated tVNS | Inhalatory-gated tVNS Then Exhalatory-gated tVNS
Started | 10 | 10
Completed | 8 | 10
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0
Period: Second Intervention (30 Minutes)
Arm/Group | Exhalatory-gated tVNS Then Inhalatory-gated tVNS | Inhalatory-gated tVNS Then Exhalatory-gated tVNS
Started | 8 | 10
Completed | 8 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exhalatory-gated tVNS Then Inhalatory-gated tVNS | Inhalatory-gated tVNS Then Exhalatory-gated tVNS | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.2 (4.9) | 30.5 (4.7) | 30.3 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 9 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Beck Depression Inventory score [Mean (Standard Deviation); unit: units on a scale] — Depression symptoms scale (minimum score =0, maximum score =63). Higher scores indicate more severe depressive symptoms. A reduction in this scale score represents an improvement in depressive symptomatology. The scale is scored by summing the ratings for each of 21 items. Each item is rated on a four-point scale ranging from 0 to 3.
  units on a scale | 30.1 (6.1) | 25.1 (8.1) | 27.3 (7.2)

OUTCOME MEASURES:

1. Primary Outcome: Brain Activity Changes (Average Differences in Beta Weights From Significantly Activated Regions: Post-stimulation Minus Pre-stimulation) Evaluated Using Functional Magnetic Resonance Imaging.
Description: A functional magnetic resonance imaging (fMRI) analysis was used to evaluate changes in brain activity [blood oxygenation level-dependent (BOLD) signal] in response to a visual stress challenge (post- and pre-stimulation). For this analysis a General Lineal Model analsysis with the statistical parametrical software (SPM) was used to model the change in BOLD signals during exposure to negative vs neutral images of the stress tasks. A voxel-wise height threshold of p < 0.001, and a cluster correction with FWE p-value<0.05 was used to identify brain areas with significant activation in response to the task. Mean beta weights within each significant cluster were extracted for each participant, and average differences in beta weights (Post minus Pre stimulation) were estimated for each group. A positive difference indicates increased activation of a particular brain region in response to the stimulation, whereas a negative difference indicates a reduction in brain activity.
Time Frame: 1 hour
Population: This is a crossover study. 20 participants were enrolled. 20 subjects completed an exhalatory-gated tVNS session and 18 and inhalatory-gated session.
Measure: Mean (Standard Deviation); unit: Beta weight difference
Arm/Group | Exhalatory-gated tVNS | Inhalatory-gated tVNS
Number analyzed (Participants) | 20 | 18
Beta weight difference
  Subgenual anterior cingulate cortex activity (Beta weight difference post-pre stimulation) | 0.60 (0.29) | -0.05 (0.12)
  Orbitofrontal cortex activity (Beta weight difference post-pre stimulation) | 0.28 (0.27) | -0.16 (0.11)
  Ventromedial prefrontal cortex activity (Beta weight difference post-pre stimulation) | 0.44 (0.38) | -0.24 (0.13)
Statistical Analysis 1: Comparison: Exhalatory-gated tVNS vs Inhalatory-gated tVNS; The null hypothesis is that there were no differences in change of brain activity in the subgenual anterior cingulate cortex (fMRI BOLD signal) between exhalatory-gated and inhalatory-gated tVNS. An ANCOVA model was used with average beta weights in response to stress task at baseline as a covariate. The test was performed with a significance level of 0.05 (two-sided); Test type: Superiority; p = 0.03, ANCOVA
Statistical Analysis 2: Comparison: Exhalatory-gated tVNS vs Inhalatory-gated tVNS; The null hypothesis is that there were no differences in change of brain activity in the orbitofrontal cortex (fMRI BOLD signal) between exhalatory-gated and inhalatory-gated tVNS. An ANCOVA model was used with average beta weights in response to stress task at baseline as a covariate. The test was performed with a significance level of 0.05 (two-sided); Test type: Superiority; p = 0.022, ANCOVA
Statistical Analysis 3: Comparison: Exhalatory-gated tVNS vs Inhalatory-gated tVNS; The null hypothesis is that there were no differences in change of brain activity in the ventromedial prefrontal cortex (fMRI BOLD signal) between exhalatory-gated and inhalatory-gated tVNS. An ANCOVA model was used with average beta weights in response to stress task at baseline as a covariate. The test was performed with a significance level of 0.05 (two-sided); Test type: Superiority; p = 0.027, ANCOVA

2. Secondary Outcome: Change in Depressive Symptoms Assessed by the Beck Depression Inventory (1 Hour Post Intervention Minus Baseline)
Description: Changes from baseline to post-stimulation in the total score of the Beck Depression Inventory (BDI) compared between exhalatory and inhalatory-gated tVNS. (Beck depression inventory minimum score= 0, maximum score= 63; higher total scores indicate more severe depressive symptoms). A positive difference at post-stimulation compared to baseline indicates an increase in depressive symptoms, whereas a negative difference indicates a reduction in depressive symptomatology.
Time Frame: 2 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Difference in BDI scale score
Arm/Group | Exhalatory-gated tVNS | Inhalatory-gated tVNS
Number analyzed (Participants) | 20 | 18
Difference in BDI scale score | -8.21 (7.4) | -3.58 (4.83)
Statistical Analysis 1: Comparison: Exhalatory-gated tVNS vs Inhalatory-gated tVNS; Null hypothesis is that there was no difference in the change in BDI scale score between exhalatory-gated tVNS and inhalatory-gated tVNS. A repeated measures ANOVA controlled by baseline values was used to test this difference. A p<0.05 was designated for statistical significance. A positive difference indicates an increase in depressive symptomatology, whereas a negative difference indicates a reduction in depressive symptoms; Test type: Superiority; p = 0.03, ANOVA

3. Secondary Outcome: Changes in Cardiac Autonomic Function (Percent Change in Normalized High-frequency Power of Heart Rate Variability (HFn-HRV): Post-stimulation Versus Pre-stimulation)
Description: Cardiac pulsatility data was collected during exposure to visual stress tasks pre- and post-stimulation and were used to estimate inter-beat intervals. A point process algorithm was then used to analyze the inter-beat intervals and evaluate heart rate variability (HRV) by separating its dynamics in the classic spectral components within the high-frequency (HF) and low-frequency (LF) ranges. Differences in normalized HF [HFn= (HF/(LF + HF))] were estimated during exposure to negative images in the fMRI stress task as a metric of parasympathetic cardiac regulation. Percent change in HFn-HRV values (Post vs Pre stimulation) were calculated for each intervention group. A positive percent change value indicates an increase in cardiovagal activity, whereas a negative change indicates a reduction in cardiovagal activity.
Time Frame: 1 hour
Population: This is a crossover study that enrolled 20 participants. HRV data from four subjects were excluded due to low-quality cardiac pulsatility signals. Thus, the HRV-related analyses were performed on data from 16 exhalatory-gated and and 16 inhalatory-gated tVNS sessions.
Measure: Mean (Standard Deviation); unit: Percent change in HF normalized units
Arm/Group | Exhalatory-gated tVNS | Inhalatory-gated tVNS
Number analyzed (Participants) | 16 | 16
Percent change in HF normalized units | 28.1 (33.9) | -0.31 (24.1)
Statistical Analysis 1: Comparison: Exhalatory-gated tVNS vs Inhalatory-gated tVNS; The null hypothesis is that there were no differences in percent HFn changes post-pre stimulation between exhalatory-gated and inhalatory-gated tVNS. A General Linear Model (GLM) analysis adjusted by baseline values was used for evaluating differences in this measure between treatment groups. A p<0.05 was designated for statistical significance. A positive percent change value indicates an increase in cardiovagal activity, whereas a negative change indicates a reduction in cardiovagal activity; Test type: Superiority; p = 0.01, Regression, Linear

ADVERSE EVENTS:
Time Frame: 1 week for each intervention (from the day of the study visit where the participants received each intervention)
Description: This is a crossover study. 20 participants were enrolled. 20 subjects completed an exhalatory-gated tVNS session and 18 and inhalatory-gated session.
Arm/Group | Exhalatory-gated tVNS | Inhalatory-gated tVNS
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/18
Other Adverse Events (participants affected / at risk) | 0/20 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-09-05): https://cdn.clinicaltrials.gov/large-docs/64/NCT04467164/Prot_SAP_000.pdf
  • Informed Consent Form (2017-07-11): https://cdn.clinicaltrials.gov/large-docs/64/NCT04467164/ICF_001.pdf